CLINICAL TRIAL: NCT04518007
Title: Hyperbaric Oxygen Therapy for Chronic Unremitting Post-Traumatic Stress Disorder (PTSD): a Prospective, Randomized, Double Blind Study
Brief Title: Hyperbaric Oxygen Therapy for Post Traumatic Stress Disorder
Acronym: HBOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 291-19
Record Dates: First submitted 2020-03-12; First posted 2020-08-19 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Post Traumatic Stress Disorder
Keywords: hyperbaric oxygen therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: hyperbaric oxygen therapy (2ATA, 100% oxygen) vs. sham (1.1ATA, 21% oxygen)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- hyperbaric oxygen therapy (HBOT) active treatment (Active Comparator): The HBOT protocol consists of 60 daily sessions, five times per week, each session lasting 90 minutes, of 100% oxygen at 2 ATA and 5-minute air breaks every 20 minutes.
  Interventions: Device: hyperbaric oxygen therapy
- hyperbaric oxygen therapy (HBOT) sham treatment (Sham Comparator): All the conditions provided in the HBOT intervention will be provided in the sham intervention. However, in contrast to the HBOT, where the pressure will go up to 2 ATA, in the sham condition the pressure will go up to 1.1 ATA during the first five minutes of the session with noise of circulating air, and then decrease slowly during the next half hour to 1.0 ATA and the oxygen level will be 21% The initial 1.1 ATA level will provide a minimal pressure sensation in the ears, with the same nurse advice on pumping the ears. In the last five minutes of the session, the air will be circulated again with its related noises. Sham and HBOT sessions will never be adjacent, so subjects from the two groups cannot meet and discuss the session and its effects.
  Interventions: Device: hyperbaric oxygen therapy

INTERVENTIONS:
Device: hyperbaric oxygen therapy — The HBOT protocol consists of 60 daily sessions, five times per week, each session lasting 90 minutes.
  Investigational product:
  Multiplace hyperbaric oxygen chamber (Haux, Germany) located at the Sago l Center for Hyperbaric Medicine and Research, Shamir (Assaf-Harofeh) Medical Center, Israel.

SUMMARY:
The study evaluates the effect of hyperbaric oxygen therapy on veterans with combat-associated PTSD in an double blind sham control study.

DETAILED DESCRIPTION:
Post-traumatic stress disorder (PTSD) is the brain's long-term imprint of a traumatic event. PTSD is characterized by intrusive thoughts, nightmares and flashbacks of past traumatic events, avoidance of trauma reminders, hypervigilance, and sleep disturbance, all of which lead to considerable social, occupational, and interpersonal dysfunction. The current available treatments for PTSD include medications and psychotherapy. However, a substantial proportion of patients have treatment resistant PTSD.

In recent years there is growing evidence that traumatic events can induce changes in the brain's structure and function that may persist months or even years after the acute event. The "non-healing brain wound" can be visualized using functional imaging. The new insight regarding the biological nature of PTSD obligates biological intervention that can induce neuroplasticity and recovery of the damage brain tissue.

Hyperbaric Oxygen Therapy (HBOT) includes the inhalation of 100% oxygen in a pressurized chamber with pressures exceeding 1 atmosphere absolute (ATA), thus enhancing the amount of oxygen dissolved in the body's tissues. It is now understood that the combined action of both hyperoxia and hyperbaric pressure together with, oxygen fluctuations generated by a pre-defined protocol may target both oxygen and pressure sensitive genes, resulting in improved mitochondrial metabolism with anti-apoptotic and anti-inflammatory effects. Moreover, these genes induce the proliferation of stem cells, augmented circulating levels of endothelial progenitor cells (EPCs) and angiogenesis factors, which induce angiogenesis and improved blood flow in the ischemic area. In recent years there is growing evidence that HBOT induced brain neuroplasticity leads to repair of chronically impaired brain functions in post-stroke and in traumatic brain injury (TBI) patients with prolonged post-concussion syndrome, even years after the brain insult, as well as in healthy aging adults. HBOT can also induce neuroplasticity and significantly improve the clinical symptoms of the most common prototype of central sensitization syndrome - fibromyalgia syndrome.

The effects of HBOT on patients suffering from chronic unremitting PTSD due to combat trauma were evaluated in a pilot study done in the investigator's institute. The recently done study included veterans with combat associated PTSD according to the Ministry of Defense (MOD) criteria, who failed to improve using the current available treatments. The results of the study demonstrated the beneficial effect of HBOT in this unfortunate severely injured unremitting PTSD population. Clinically significant improvement was demonstrated in a major fraction of study participants. In correlation with the clinical improvement, a significant improvement in brain activity was demonstrated in the functional MRI imaging.

The aim of the current study is to evaluate the effect of HBOT on chronic unremitting combat associated PTSD in an double blind sham control study

ELIGIBILITY:
Inclusion Criteria:

* Subject willing and able to read, understand and sign an informed consent
* Age 25-60
* Five years or more after the last traumatic exposure
* CAPS-5 score PTSD symptoms questionnaire ≥ 20.
* Failure to improve after at least one line of conventional therapy, such as prolonged exposure, trauma related psychotherapy, eye movement desensitization therapy (EMDR).
* Stable psychological and pharmacological treatment for more than three months prior to inclusion.

Exclusion Criteria:

* Inability to attend scheduled clinic visits and/or comply with the study protocol.
* History of TBI or any other brain pathology
* Active malignancy
* Substance use at baseline, except for prescribed cannabis if vaporized or taken PO as tincture
* Current manic episode or psychotic disorders
* Serious suicidal ideation
* Severe or unstable physical disorders or major cognitive deficits at baseline
* for any reason prior to study enrollment
* Chest pathology incompatible with pressure changes (including active asthma)
* Ear or Sinus pathology incompatible with pressure changes
* An inability to perform an awake brain MRI
* active smoking

Ages: 25 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
PTSD symptoms | Change from Baseline immediately after the intervention
  PTSD symptoms will be assessed by the PTSD Clinician-Administered PTSD Scale (CAPS) questionnaire.

SECONDARY OUTCOMES:
depression | Change from Baseline immediately after the intervention
  Beck depression inventory II
Changes in growth following a traumatic event | Change from Baseline immediately after the intervention
  The post-traumatic growth inventory (PTGI)
wellbeing | Change from Baseline immediately after the intervention
  Changes will be measured by the wellbeing inventory (WBI).
emotional regulation | Change from Baseline immediately after the intervention
  Changes in emotional regulation will be measured by the emotion regulation questionnaire (ERQ).
global distress | Change from Baseline immediately after the intervention
  The brief symptom inventory (BSI)
sleep quality | Change from Baseline immediately after the intervention
  Changes in sleep patterns will be measured using the Pittsburgh sleep quality index (PSQI).
Depression, anxiety and stress | Change from Baseline immediately after the intervention
  Depression, anxiety and stress will be evaluated using scale-21 items (DASS-21)
Daily documentation of symptoms | daily during intervention, up to 16 weeks
  Daily distress and change in symptoms will be evaluated using visual assessment scale (VAS) based questionnaire
Mind streams cognitive health assessment (Mind streams) | Change from Baseline immediately after the intervention
  memory, attention and information process will be evaluated using the Mind streams cognitive health assessment (Mind streams)
MRI Imaging | Change from Baseline immediately after the intervention
  At each of the evaluations, patients will undergo structural and functional MRI scanning. Images will be acquired on Vida 3 Tesla Scanner, configured with a 64-channel receiver head coils (Siemens Healthcare, Erlangen, Germany) at Shamir medical center radiology department.
Brain SPECT | Change from Baseline immediately after the intervention
  SPECT will be conducted with 925-1,110 (25-30 mCi) of technetium-99m-methyl-cysteinate-dimmer (Tc-99m-ECD) at 40-60 min post injection, using a dual detector gamma camera (Siemens Medical Systems) equipped with high resolution collimators
Cardiopulmonary exercise test | Change from Baseline immediately after the intervention
  The cardiopulmonary exercise test (CPET) is a noninvasive measurement of the cardiovascular system, respiratory system and muscles
Immune system | Change from Baseline immediately after the intervention
  Inflammatory cytokines: blood tests will include: interleukin (IL) IL-1, IL-6, tumor necrosis factor-alpha, C reactive protein and T cells panel

CONTACTS AND LOCATIONS:
Overall Officials: Keren Doenyas, Principal Investigator — Asaf-Harofhe MC
Locations (1):
- Dialysis Clinic in Asaf Harofhe Medical Center, Ẕerifin, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Danan D, Grosskopf Y, Mayo A, Efrati S, Kutz I, Lang E, Alon U, Doenyas-Barak K. Hyperbaric Oxygen Therapy for PTSD: Threshold Effect for Sustained Symptom Improvement in a Biologically Based Treatment. Brain Behav. 2025 Aug;15(8):e70757. doi: 10.1002/brb3.70757. PMID 40847457
- [Derived] Doenyas-Barak K, Kutz I, Lang E, Assouline A, Hadanny A, Aberg KC, Levi G, Beberashvili I, Mayo A, Efrati S. Hyperbaric Oxygen Therapy for Veterans With Combat-Associated Posttraumatic Stress Disorder: A Randomized, Sham-Controlled Clinical Trial. J Clin Psychiatry. 2024 Nov 10;85(4):24m15464. doi: 10.4088/JCP.24m15464. PMID 39566051